CLINICAL TRIAL: NCT02247284
Title: Study to Investigate Reproducibility of the New Heidelberg Spectralis SD-OCT Glaucoma Module Premium Edition (Software Version 6.0) in Comparison to Reproducibility of RNFL Scans.
Brief Title: Reproducibility of RNFL and ONH Measurements in OAG With Heidelberg Spectralis SD-OCT Glaucoma Module Premium Edition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Glaucoma-Premium-OCT
Record Dates: First submitted 2014-09-16; First posted 2014-09-25 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- group 1 (Experimental): patient with a diagnosis of primary open angle glaucoma will undergo 'RNFL and BMO-MRW SD-OCT' measurements with Heidelberg Spectralis SD-OCT old protocoll and Glaucoma Premium Module (new) protocoll, which in addition to RNFL measurements include measurement of Bruch's Membrane Opening-based minimum rim width (BMO-MRW).
  Interventions: Device: RNFL and BMO-MRW SD-OCT

INTERVENTIONS:
Device: RNFL and BMO-MRW SD-OCT — Masurement of peripapillary RNFL measurements with Heidelberg Spectralis SD-OCT (Heidelberg Engeneering GmbH, Heidelberg, Germany) old protocoll and in addition with the new Glaucoma Premium Module (software version 6.0) tocoll, which in addition to RNFL measurements include measurement of Bruch's Membrane Opening-based minimum rim width (BMO-MRW).

SUMMARY:
The purpose of this study is to assess and compare the repeatability of SD-OCT (Spectralis™ OCT, Version 6.0, Heidelberg Engineering, Germany) RNFL thickness measurements with a new software (glaucoma premium module) with the well established peripapillary RNFL thickness measurements in patients with primary open angle glaucoma.

DETAILED DESCRIPTION:
The purpose of this study is to assess and compare the repeatability of SD-OCT (Spectralis™ OCT, Version 6.0, Heidelberg Engineering, Germany) RNFL thickness measurements with the new software (method B) and with the previous method of measurement (method A) in patients with glaucoma.

It is a prospective, not blinded, not randomised, monocentric study. Inclusion of 50 patients with a diagnosis of primary open angle glaucoma (POAG), that will be recruited from the ophthalmology outpatient department of the UniversityHospital Zurich, Switzerland. All patients will undergo a full ophthalmic examination including measurement of refraction, best corrected visual acuity, examination of anterior and posterior compartment and measurement of the intraocular pressure. On the same day they will have 3 OCT examinations with a new method of measurement (method B).On the same day the first 10 patients will undergo also 3 OCT examinations with the previous method (method A) and they will get an other 3 OCT examinations with method B by a second observer. For this 10 patients the next consultation (3 months +/- 1 month) the 3 OCT examinations with method B will be repeated by the first observer.

Primary objectives are coefficient of variations (COV) of method A and B; Intra-class-correlations (ICC) of method A and B.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of POAG glaucoma
* male and female patients aged 18 years or older, no upper limit
* written informed consent
* visual acuity of more or equal to 0.5 Snellen
* refractive error between + /- 6.00 D spheric and under or equal than 2.00 D cylindrical

Exclusion Criteria:

* history of surgery other than uncomplicated cataract surgery
* disease affecting cornea, anterior compartment, lens, vitreous body
* history of severe ocular disease, particularly diseases affecting the optic nerve, other than glaucoma
* history of ocular trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Retinal nerve fiber layer thickness (RNFL) | baseline and 3 months +/- 1 month
  Retinal nerve fiber layer thickness (RNFL) measured with Spectralis OCT
Bruch's membrane opening-based minimum rim width (BMO-MRW) | baseline and 3 months +/- 1 month
  Bruch's membrane opening-based minimum rim width (BMO-MRW) measured with Spectralis OCT

SECONDARY OUTCOMES:
Coefficient of variations (COV) of RNFL and BMO-MRW | baseline and 3 months +/- 1 month
  Coefficient of variations (COV) of RNFL and BMO-MRW
Intra-class-correlations (ICC) of RNFL and BMO-MRW | baseline and 3 months +/- 1 month
  Intra-class-correlations (ICC) of RNFL and BMO-MRW

CONTACTS AND LOCATIONS:
Overall Officials: Jens Funk, MD, PhD, Principal Investigator — UniversityHospital Zurich, Zurich, Switzerland
Locations (1):
- UniversityHospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No